CLINICAL TRIAL: NCT04970810
Title: My Diabetes, My Community
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: IRB20-0870; 1R01DK127961-01 (NIH)
Record Dates: First submitted 2020-05-18; First posted 2021-07-21 (Actual); Results first posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-10

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant
Masking Description: This will be a single-blind study, and subjects will blinded to the different group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Attention Control (No Intervention): Subjects monthly calls similar in structure to the intervention arms, but without support. (attention placebo control)
- My Diabetes Goal (Active Comparator): My Diabetes Goal protocol
  Interventions: Behavioral: My Diabetes Goal
- My Diabetes Goal + Community Rx (Active Comparator): My Diabetes Goal protocol + Community Rx protocol
  Interventions: Behavioral: My Diabetes Goal + CommunityRx

INTERVENTIONS:
Behavioral: My Diabetes Goal — Subjects enrolled in the MDG arm will receive surveys at baseline, 6 months and 12 months, followed by monthly diabetes care management phone calls.
  Arms: My Diabetes Goal
Behavioral: My Diabetes Goal + CommunityRx — Subjects enrolled in the MDG arm + CRx will receive surveys at baseline, 6 months and 12 months, followed by monthly diabetes care management phone calls. Participants will also receive a HealtheRx (personalized resource "prescriptions") for community organizations.
  Arms: My Diabetes Goal + Community Rx

SUMMARY:
Older adults with diabetes are a highly vulnerable population that suffers the highest rates of cardiovascular and microvascular complications as well as adverse drug events such as hypoglycemia. Investigators will conduct a 12-month pragmatic clinical trial evaluating the impact of scalable interventions that are designed to support personalized goal setting and self-care through remote delivery of clinical and socioeconomic risk assessment, telephonic care management, and community resource linkage. This highly personalized approach to diabetes care has to potential to improve quality of life of this high-risk population while avoiding adverse drug events.

DETAILED DESCRIPTION:
To address the needs of older patients with diabetes, multiple organizations have called for a personalized approach to setting risk factor goals and self-care plans. The American Geriatrics Society (AGS) and the American Diabetes Association (ADA) have published recommendations urging individualized glycemic goals (hemoglobin A1C (A1C) <7.5%, <8.0%, or <8.5%) for three strata of older patients (healthy, complex, very complex). The guidelines also acknowledge the importance of addressing socioeconomic risks that are barriers to self-care management such as cost-related non-adherence and food insecurity. Despite widespread agreement by experts, the clinical impact of this highly personalized approach to diabetes care for older adults has been rarely studied in controlled trials. Interventions designed to personalize diabetes care must overcome multiple challenges to implementation including the brief clinical encounter, lack of patient engagement between encounters, and lack of systems to leverage community-based self-care resources.

Investigators propose to address these knowledge and care gaps by studying the integration of two evidence-based interventions designed to engage patients and enhance self-care:. Managing Diabetes to Gain Opportunities for a More Active Life (My Diabetes GOAL) and CommunityRx. The My Diabetes GOAL intervention is designed to engage older patients in personalized goal setting and chronic disease management.

ELIGIBILITY:
Inclusion Criteria:

1. History of type 2 diabetes
2. Seen in clinic within past year
3. A1C>7.5%
4. Community dwelling
5. Access to personal email address OR internet access
6. Speaks and reads English
7. Resides in the target geographic region (zip codes)

Exclusion Criteria:

1. Unable to consent to study for themselves
2. Prior participation in CRxCaregiver, CRxHunger, or My Diabetes GOAL trials

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 512 (Actual)
Dates: Start 2021-07-29 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2024-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elbert Huang, Principal Investigator — University of Chicago; Stacy Lindau, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago Medicine, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No
We do not plan to share IPD with other researchers.

REFERENCES:
- [Derived] Abramsohn EM, De Ornelas M, Borson S, Frazier CR, Fuller CM, Grana M, Huang ES, Jagai JS, Makelarski JA, Miller D, Schulman-Green D, Shiu E, Thompson K, Winslow V, Wroblewski K, Lindau ST. Two concurrent randomized controlled trials of CommunityRx, a social care intervention for family and friend caregivers delivered at the point of care. Res Sq [Preprint]. 2023 Mar 1:rs.3.rs-2464681. doi: 10.21203/rs.3.rs-2464681/v1. PMID 36909590

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Attention Control | My Diabetes Goal | My Diabetes Goal + Community Rx
Started | 170 | 173 | 169
Completed 6 Month Follow up Survey | 156 | 152 | 149
Completed 12 Month Follow-up Survey | 156 | 146 | 147
Completed | 167 | 173 | 165
Not Completed | 3 | 0 | 4
Not completed — deemed ineligible after randomization | 3 | 0 | 4

BASELINE CHARACTERISTICS:
Population: Does not include 7 deemed ineligible after randomization.
Groups:
- Total: Total of all reporting groups
Arm/Group | Attention Control | My Diabetes Goal | My Diabetes Goal + Community Rx | Total
Number analyzed (Participants) | 167 | 173 | 165 | 505
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.9 (6.3) | 68.8 (5.9) | 69.2 (6.7) | 69.0 (6.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 105 | 114 | 113 | 332
  Male | 62 | 59 | 52 | 173
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 123 | 126 | 129 | 378
  White | 28 | 33 | 25 | 86
  Other | 16 | 14 | 11 | 41
Region of Enrollment [Number; unit: participants]
  United States | 167 | 173 | 165 | 505
Most Recent A1C Value [Mean (Standard Deviation); unit: % (percentage of A1C)] | 9.0 (1.5) | 9.1 (1.6) | 9.0 (1.5) | 9.0 (1.5)
Diabetes Empowerment Scale (DES) [Mean (Standard Deviation); unit: units on a scale] — A standardized questionnaire including 28 questions with response categories of 'strongly disagree', 'somewhat disagree', 'neutral', 'somewhat agree', and 'strongly agree'. A total score for the DES is calculated by summing all of the item scores and dividing by 28 for a possible score range of 1-5, where a higher score indicates a higher level of empowerment.
  units on a scale | 4.2 (0.6) | 4.3 (0.5) | 4.1 (0.6) | 4.2 (0.6)

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Percent of Hemoglobin A1C
Description: Mean change in percent of hemoglobin A1C from baseline to month 12.
Time Frame: Baseline to 12 months
Population: There are missing 12 month A1C values for all three study arms.
Measure: Mean (Standard Deviation); unit: percentage of hemoglobin A1C
Arm/Group | Attention Control | My Diabetes Goal | My Diabetes Goal + Community Rx
Number analyzed (Participants) | 138 | 139 | 129
percentage of hemoglobin A1C | -1.1 (1.79) | -0.8 (2.1) | -0.8 (1.5)
Statistical Analysis 1: Comparison: Attention Control vs My Diabetes Goal; Test type: Superiority; p = 0.8, Mixed Models Analysis
Statistical Analysis 2: Comparison: Attention Control vs My Diabetes Goal + Community Rx; Test type: Superiority; p = 0.3, Mixed Models Analysis
Statistical Analysis 3: Comparison: My Diabetes Goal vs My Diabetes Goal + Community Rx; Test type: Superiority; p = 0.5, Mixed Models Analysis

2. Secondary Outcome: Number of Participants With Documentation of Diabetes Goal at Baseline and Month 12
Description: We reviewed the electronic health records (EHR) to assess how many participants had a documented goal in the EHR at baseline and at 12 months. The possible values will be yes or no goals documented in the EHR.
Time Frame: Baseline to 12 months
Population: The number of analyzed A1C goal results is dependent on the number of survey respondents.
Measure: Count of Participants; unit: Participants
Arm/Group | Attention Control | My Diabetes Goal | My Diabetes Goal + Community Rx
Number analyzed (Participants) | 167 | 173 | 165
Participants
  Documented Goals at Baseline | 52 | 60 | 43
  Documented Goals After Baseline: number analyzed (Participants) | 162 | 166 | 156
  Documented Goals After Baseline | 43 | 165 | 156
Statistical Analysis 1: Comparison: Attention Control vs My Diabetes Goal vs My Diabetes Goal + Community Rx; Documented goals at baseline for all three arms; Test type: Superiority; p = 0.2, Chi-squared
Statistical Analysis 2: Comparison: Attention Control vs My Diabetes Goal vs My Diabetes Goal + Community Rx; Documented goals after Baseline in all three arms; Test type: Superiority; p < 0.001, Chi-squared

3. Secondary Outcome: Personalized A1C Goals
Description: The A1C goal outcome is based on a survey response and is distinct from the measured A1C from laboratory testing. Goal setting conversation with nurse occurred during Month 1 call.
Time Frame: Baseline to Month 1 Call
Population: The number of analyzed A1C goal results is dependent on the number of survey respondents in the two intervention arms. The Attention Control arm did not include a goal setting conversation with a nurse.
Measure: Mean (Standard Deviation); unit: % (percentage A1c)
Arm/Group | My Diabetes Goal | My Diabetes Goal + Community Rx
Number analyzed (Participants) | 173 | 165
% (percentage A1c)
  Initial Goal | 6.6 (0.9) | 6.7 (0.7)
  Modified Goal: number analyzed (Participants) | 170 | 160
  Modified Goal | 7.1 (0.8) | 7.1 (0.7)
Statistical Analysis 1: Comparison: My Diabetes Goal vs My Diabetes Goal + Community Rx; Initial goal at baseline; Test type: Superiority; p = 0.7, Chi-squared
Statistical Analysis 2: Comparison: My Diabetes Goal vs My Diabetes Goal + Community Rx; Modified goal after Month 1 call with nurse; Test type: Superiority; p = 0.6, Chi-squared

4. Secondary Outcome: Number of Participants Who Achieved Personalized A1C Goals
Description: Investigators will measure whether or not patients are reaching the modified goals they have documented in the survey, among those who have set up their personalized goals. The possible values will be yes or no reaching personalized goals.
Time Frame: Baseline to 12 months
Population: The number of analyzed A1C goal results is dependent on the number of survey respondents in the two intervention arms. The Attention Control arm did not include a goal setting exercise.
Measure: Count of Participants; unit: Participants
Arm/Group | My Diabetes Goal | My Diabetes Goal + Community Rx
Number analyzed (Participants) | 170 | 160
Participants
  Achieved Goal at Baseline | 5 | 1
  Achieved Goal at 12 Months: number analyzed (Participants) | 136 | 128
  Achieved Goal at 12 Months | 38 | 34
Statistical Analysis 1: Comparison: My Diabetes Goal vs My Diabetes Goal + Community Rx; Achieved goal at baseline across three arms; Test type: Superiority; p = 0.2, Chi-squared
Statistical Analysis 2: Comparison: My Diabetes Goal vs My Diabetes Goal + Community Rx; Achieved goal at 12 months across all three arms; Test type: Superiority; p = 0.9, Chi-squared

5. Secondary Outcome: Diabetes Empowerment Scale (DES)
Description: Evaluate subject self-efficacy through the Diabetes Empowerment Scale (DES). DES is a standardized questionnaire including 28 questions with response categories of 'strongly disagree', 'somewhat disagree', 'neutral', 'somewhat agree', and 'strongly agree'. A total score for the DES is calculated by summing all of the item scores and dividing by 28 for a possible score range of 1-5 where a higher score indicates a higher level of empowerment.
Time Frame: Baseline to 12 months
Population: Number analyzed is dependent on survey respondents.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Attention Control | My Diabetes Goal | My Diabetes Goal + Community Rx
Number analyzed (Participants) | 156 | 146 | 148
score on a scale | -0.1 (1.0) | -0.2 (1.2) | 0.03 (1.1)
Statistical Analysis 1: Comparison: Attention Control vs My Diabetes Goal; Test type: Superiority; p = 0.9, Mixed Models Analysis
Statistical Analysis 2: Comparison: Attention Control vs My Diabetes Goal + Community Rx; Test type: Superiority; p = 0.2, Mixed Models Analysis
Statistical Analysis 3: Comparison: My Diabetes Goal vs My Diabetes Goal + Community Rx; Test type: Superiority; p = 0.1, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Attention Control | My Diabetes Goal | My Diabetes Goal + Community Rx
All-Cause Mortality (participants affected / at risk) | 1/167 | 3/173 | 4/165
Serious Adverse Events (participants affected / at risk) | 0/167 | 0/173 | 0/165
Other Adverse Events (participants affected / at risk) | 0/167 | 0/173 | 0/165

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-11-15): https://cdn.clinicaltrials.gov/large-docs/10/NCT04970810/Prot_SAP_001.pdf
  • Informed Consent Form (2022-12-16): https://cdn.clinicaltrials.gov/large-docs/10/NCT04970810/ICF_002.pdf